CLINICAL TRIAL: NCT03534219
Title: Efficacy of the EarPopper Device in Children With Recurrent Otitis Media: A Randomized Controlled Trial
Brief Title: Efficacy of the EarPopper Device in Children With Recurrent Otitis Media
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Tristan Tham, Research Scientist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-0388-LHH
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Recurrent Acute Otitis Media; Acute Otitis Media
Keywords: Earpopper; Prophylaxis; Randomized controlled trial
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized in a 1:1 ratio using permuted blocks. Subjects will be stratified by site (Lenox Hill) prior to randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since there will be no dummy devices in this trial, we will be unable to blind the patients and physicians to whom is using the EP device. The assessors/data collectors will be blinded for patient follow-up, and the statistician will be blinded. Therefore this will be a double blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Arm: EarPopper (Experimental): All patients in this arm will receive the EarPopper device.
  Length of administration: 1 year Dose: Dosing of the EP device will be twice per day, once in the morning and once before bedtime. This is consistent with previous dosing which showed no adverse events and an excellent safety profile. 5, 6
  Administration:
  1. Hold nosepiece firmly against nostril opening creating a good, tight seal is crucial. Plug the other nostril closed.
  2. Push button to start the airflow and swallow while the device is running.
  3. Repeat on other nostril. After 5 minutes, repeat steps 1 - 3. This will complete one treatment.
  Telephone call survey:
  Will be administered monthly by study investigator. Telephone call survey is based on the OMO-22 Form.
  Interventions: Device: EarPopper
- Control (No Intervention): All patients in this arm will not receive any intervention. EarPopper device will be given to this group at the end of follow-up period (1 year)
  Telephone call survey:
  Will be administered monthly by study investigator. Telephone call survey is based on the OMO-22 Form.

INTERVENTIONS:
Device: EarPopper — The EP device is 510(K) regulated (510(K) Number K073401) as a non-surgical, non-drug related treatment for middle ear pressure problems. The device is based on the Politzer Maneuver, and works by opening the Eustachian tube by delivering a safe, constant stream of air into the nasal cavity. In clinical studies funded by the National Institutes of Health (Grant#: 5R44DC003613-03), the EarPopper has proven to be effective in reducing chronic middle ear effusions. By regularly aerating the middle ear, we hypothesize that the EarPopper device will be an effective prophylactic measure to reduce incidence of AOM in children with recurrent OM. The device delivers a jet of air pressure from the nozzle at 5.2PSI, at a volume velocity of 1,524mL/min.
  Arms: Intervention Arm: EarPopper

SUMMARY:
This is a randomized controlled clinical trial evaluating the efficacy of the EarPopper device (EP) in the reduction of episodes of acute otitis media (AOM) in children with recurrent otitis media. The control arm will be observational. The intervention arm will have the EP used.

DETAILED DESCRIPTION:
The hypothesis of this randomized controlled trial is that the EP device will be able to prophylactically decrease incidence of AOM in children with recurrent AOM. The secondary hypothesis is that the EP device will be able to decrease morbidity of AOM and severity of AOM in children with recurrent AOM (by measuring quality of life and associated endpoints).

The EP device is 510(K) regulated (510(K) Number K073401) as a non-surgical, non-drug related treatment for middle ear pressure problems such as: Middle ear fluid (Otitis Media with Effusion), Eustachian Tube Dysfunction, Temporary hearing loss, Ear pain and pressure caused by air travel, Ear fullness caused by colds, allergies and sinusitis.

This is a randomized, controlled, double blinded study. This is a randomized controlled clinical trial evaluating the efficacy of the EarPopper device (EP) in the reduction of episodes of acute otitis media (AOM) in children with recurrent otitis media. The control arm will be observational.

Patients will be followed up for a period of one year, and monthly telephone call interviews will be conducted.

All patients will receive the EarPopper device for participation in this trial (for the control arm, they will receive the device at the end of their study follow up).

ELIGIBILITY:
INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form from parent, plus assent form (if age appropriate)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 4-11
4. Diagnosed with recurrent AOM, defined as: least 2 episodes of AOM within the preceding year of date of screening
5. Must be able to follow directions to use EarPopper, or have a caregiver able to administer the device.
6. Patient must be currently free of middle ear effusion or current acute OM. This will be determined on physical examination during screening visit

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patient with chronic middle ear effusion.
2. Patients with potential complications or confounding conditions: asthma, chronic sinusitis, immunodeficiency, diabetes mellitus
3. Patient with cleft palate.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AOM | 1 year
  Null Hypothesis: The incidence of AOM is the same between two arms of the study. Description: Definition of AOM will be presence of AOM documented in the clinic notes during the follow-up period. This is a binary data point.
  Test: chi-square test with a 0.05 two-sided significance level

SECONDARY OUTCOMES:
Hazard ratio of time to AOM | 1 year
  Null hypothesis: Hazard ratios between groups is the same. Test: Cox proportional hazards ratio (CPH) model for time-to-event data will be computed. Actuarial data will be displayed as Kaplan Meier curves (KM) and the differences between the curves will be tested with the Log-rank test. Assumptions for proportional hazards will be conducted to ensure that the data obtained fulfills the criteria for the Cox model.
Proportion of patients without AOM and antibiotics use | 1 year
  Null hypothesis: Proportion is the same between groups. Test: Fisher exact test will be used to compare the proportions
Otitis Media Outcome-22 (OMO-22) form and questionnaire | 1 year
  Null hypothesis: Otitis Media Outcome-22 form scores are the same between the two arms of the study.
  Description: The Otitis Media Outcome-22 form is a 22-item questionnaire based on a 7-point Likert scale. The questionnaire is divided into physical, emotional, hearing loss, speech, and social symptoms subsets. The Likert range is 0-6, 0 being no problem and 6 being the worst.
  The total score is calculated by adding up all the scores from the 22 individual questions. Therefore, the max possible total score is = (6 for each individual item) * (22 items) = 132. Range of total score = 0-132. The higher the total score, the worse the impact of otitis media in the patient.
  Test: Significance testing between timepoints will be performed using paired t test statistics for parametric data with equal distributions and the Mann-Whitney rank sum test for nonparametric data.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Tham, MD, Principal Investigator — Lenox Hill Hospital
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Sharing plan is currently undecided

REFERENCES:
- [Background] Arick DS, Silman S. Nonsurgical home treatment of middle ear effusion and associated hearing loss in children. Part I: clinical trial. Ear Nose Throat J. 2005 Sep;84(9):567-8, 570-4, 576 passim. PMID 16261757
- [Background] Silman S, Arick DS, Emmer MB. Nonsurgical home treatment of middle ear effusion and associated hearing loss in children. Part II: Validation study. Ear Nose Throat J. 2005 Oct;84(10):646, 648, 650 passim. PMID 16382747
- [Background] Banigo A, Hunt A, Rourke T, Whiteside O, Aldren C. Does the EarPopper((R)) device improve hearing outcomes in children with persistent otitis media with effusion? A randomised single-blinded controlled trial. Clin Otolaryngol. 2016 Feb;41(1):59-65. doi: 10.1111/coa.12480. PMID 26095773